CLINICAL TRIAL: NCT00097370
Title: An Open Label Extension Study to Evaluate Safety and Efficacy of Mepolizumab in Patients With Hypereosinophilic Syndromes
Brief Title: Open-Label Extension Of Intravenous Mepolizumab In Patients With Hypereosinophilic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor (29 Sep 2010). Subjects eligible to continue mepolizumab treatment were transferred into the compassionate use program (MHE104317)
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100901
Record Dates: First submitted 2004-11-22; First posted 2004-11-23 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Mepolizumab; Open-label; Anti-IL-5; Hypereosinophilic Syndrome; Hypereosinophilia
MeSH Terms: conditions — Hypereosinophilic Syndrome; Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mepolizumab (Experimental): 750mg Intravenous, monthly and individual dosing schedule
  Interventions: Drug: mepolizumab

INTERVENTIONS:
Drug: mepolizumab — Study Drug

SUMMARY:
This is an open label study of mepolizumab 750 mg intravenous in those subjects who participated in study 100185 to evaluate the long term safety and efficacy of mepolizumab in subjects with hypereosinophilic syndrome. The study will also evaluate the optimal dosing frequency for clinical use, the effects on corticosteroid reduction, and decrease of signs and symptoms of Hypereosinophilic Syndrome.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent.
* Subjects who have participated in Study MHE100185 and have been administered at least 2 doses of study medication.
* Not pregnant or nursing
* Of non-childbearing potential (i.e., women who had a hysterectomy, are post-menopausal which is defined as 1 year without menses, have both ovaries surgically removed, or have current documented tubule ligation); or
* Of childbearing potential (i.e., women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea [even severe], women who are perimenopausal or have just begun to menstruate. These women must have a negative serum pregnancy test at the Screening Visit, and agree to one of the following:1). Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of investigational product until 3 months after the last dose of investigational product; Or 2). Consistent and correct use of one of the following acceptable methods of birth control for one month prior to the start of the investigation product and three months after the last dose:Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subjects; Implants of levonorgestrel;Injectable progestogen;Any intrauterine device (IUD) with a documented failure rate of less than 1% per year; Oral contraceptives (either combined or progestogen only)

Exclusion criteria:

* Has developed life-threatening or other serious illness or clinical manifestation deemed inappropriate for inclusion in study per the principal investigator
* Has any of the following abnormal laboratory values at the Week36/EW Visit of Study MHE100185: • Serum creatinine ≥3 times institutional upper limit normal (ULN); • AST or/ALT ≥5 times institutional ULN; • Platelet count < 50,000/uL
* Has developed abnormal cardiac functions, as the following, within past 3 months:• Left ventricular ejection fraction (LVEF) < 20%; • NYHA class IIIb or IV; • Angina or acute myocardial infarction
* Has developed allergic reaction to Study MHE100185 investigational product Use of an investigational drug as concurrent medication
* Does not complete Week36/EW Visit assessments required in Study MHE100185
* Has completed or been terminated from Study MHE100185 for more than 1 month
* Recent history or suspicion of current drug abuse or alcohol abuse within the last 6 months
* Positive pregnancy test at the Week36/EW Visit of Study MHE100185

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2010-09-29 (Actual); Study Completion 2010-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (10):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Australia (2):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, West Perth, Western Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (4):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
- France (2):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Suresnes
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
- GSK Investigational Site, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 100901 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) who completed 9 months of treatment or withdrew from Study MHE100185 after receiving >=2 infusions of study medication were enrolled in this open label extension study. Par. with daily dose of prednisone >10 milligrams (mg) or <=10 mg at the end of Study MHE100185 were enrolled in Stage 1 or Stage 2 of this study, respectively.
Pre-assignment Details: This study was open-label extension to previous Study MHE100185 (NCT00086658). A total of seventy-eight participants participated in this study. Of these, 38 participants previously received placebo in Study MHE100185 and 40 participants previously received mepolizumab in Study MHE100185.
Groups:
- Mepolizumab 750 mg: Participants received mepolizumab 750 mg by intravenous (IV) infusion monthly in Stage 1 along with concomitant hypereosinophilic syndrome (HES)-active medications that included prednisone (or equivalent) or other HES therapies. In Stage 2, the dosing intervals were optimized for each participant based on the individual's blood eosinophil count and the clinical presentation. In Stage 3, the dosing frequency established in Stage 2 was continued with individual participant monitoring.
Period: Stage 1
Arm/Group | Mepolizumab 750 mg
Started | 37 (Participants entered from study MHE100185.)
Completed | 31
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 2
Period: Stage 2
Arm/Group | Mepolizumab 750 mg
Started | 72 (41 participants entered from study MHE100185 and 31 participants continued from Stage 1.)
Completed | 59
Not Completed | 13
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 3
Not completed — Pregnancy | 1
Not completed — Sponsor Terminated Study | 2
Not completed — Lost to Follow-up | 1
Period: Stage 3
Arm/Group | Mepolizumab 750 mg
Started | 59 (Participants continued from Stage 2.)
Completed | 0
Not Completed | 59
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 1
Not completed — Sponsor Terminated Study | 52
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Mepolizumab 750 mg: Participants received mepolizumab 750 mg by IV infusion monthly in Stage 1 along with concomitant HES-active medications that included prednisone (or equivalent) or other HES therapies. In Stage 2, the dosing intervals were optimized for each participant based on the individual's blood eosinophil count and the clinical presentation. In Stage 3, the dosing frequency established in Stage 2 was continued with individual participant monitoring.
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  Arabic/North African | 2
  Black | 6
  East and South East Asian | 2
  South Asian | 1
  White/Caucasian | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) During the Treatment Phase
Description: An AE is any untoward medical occurrence in clinical investigation participants temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs are summarized by Treatment phase. Safety and tolerability of the study drug was assessed by number of participants with any AE
Time Frame: From the first dose of study medication up to 7 days after the last dose (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population: all enrolled participants who received at least one dose of mepolizumab in this study.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Participants | 76

2. Primary Outcome: Number of Participants With Any Adverse Event (AE) During the Follow-up Phase
Description: An AE is any untoward medical occurrence in clinical investigation participants temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs are summarized by Follow-up phase. Safety and tolerability of the study drug was assessed by number of participants with any AE
Time Frame: From end of Treatment Phase up to 97 days after the last dose date (up to approximately 6 years)
Population: Follow-up Population: subset of the modified ITT Population who had evidence of being in the study > length of dosing cycle + 7 days after the date of their last dose of study medication and up to and including 97 days after their last dose date.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 15
Participants | 3

3. Secondary Outcome: Number of Participants Achieving a Prednisone Level of =<10 mg (as Sole Background Therapy) at the End of Study
Description: Participants who were receiving a prednisone dose level of =<10 mg as their sole background therapy at the end of the study were included for the analysis.
Time Frame: up to approximately 6 years
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Participants | 62

4. Secondary Outcome: Number of Participants Achieving an Eosinophil Level of < 600 Cell/Microliter (uL) (in Addition to the Lowest Background Therapy) at the End of Study
Description: The criteria for eosinophil count was achieved if the participant's eosinophil count remained below <600 cell/uL for the last observation on study i.e. within length of dosing cycle + 7 days of last dose of study drug. For participants who entered in Stage 1, HES medications taking prior to the first infusion date in Stage 2 were considered as the lowest background therapy. For participants who entered in Stage 2, HES medications taken on the date that immediately preceded the first infusion date of study drug and had not been discontinued was regarded as the lowest background therapy. If the dose of the lowest background therapy had increased or the medication had changed or the participant had not reached their lowest background therapy, the participant was regarded as not achieving this endpoint.
Time Frame: up to approximately 6 years
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Participants | 46

5. Secondary Outcome: For Those Participants Who Completed 9 Months of Dosing in Study MHE100185 and Achieved a Prednisone Level <=10 mg: Number of Participants Achieving <= 10 mg Prednisone (as Sole Background Therapy) for >= 3months
Description: Participants from study MHE100185 who completed the 9 months treatment period and achieved a level of <=10 mg of prednisone at study end were analyzed. Duration of doses <=10 mg was determined by examining changes in the prednisone dosing or allowable alternative corticosteroid medication (prednisone equivalents). Start and stop dates of other HES medications were checked to ensure that they did not overlap with the steroid dosing dates. If it did, then the number of days <=10 mg during this overlap was considered as zero and the cumulative days reset to zero, as the endpoint was assessing prednisone dose as sole background therapy. The dosing criteria for this endpoint was considered as achieved if the duration of dosing was minimum of 84 days (3months).
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants who completed 9 months of dosing in study MHE100185 and achieved a prednisone level <=10 mg were analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 43
Participants | 39

6. Secondary Outcome: For Those Participants Who Completed 9 Months of Dosing in Study MHE100185 and Achieved a Prednisone Level >10 mg: Number of Participants Achieving <=10 mg Prednisone (as Sole Background Therapy) for >= 8 Weeks
Description: Participants from study MHE100185 who completed the 9 months treatment period and achieved a level of prednisone of >10 mg at the end of the study were analyzed. Duration of doses <= 10 mg were determined by examining changes in the prednisone dosing or allowable alternative corticosteroid medication (prednisone equivalents). Start and stop dates of other HES medications were checked to ensure that they did not overlap with the steroid dosing dates. If overap occurred, then the number of days <=10 mg during this overlap was considered as zero and the cumulative days reset to zero, as the endpoint was assessing prednisone dose as sole background therapy. The dosing criteria for this endpoint was considered as achieved if the duration of dosing was minimum of 53 days (8 weeks).
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants who completed 9 months of dosing in study MHE100185 and achieved a prednisone level >10 mg were analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 6
Participants | 5

7. Secondary Outcome: For Those Participants Who Entered Stage 2 From Study MHE100185 With a Prednisone Level of <=10 mg Prednisone: Number of Participants Achieving a Prednisone Dose <=10 mg (as Sole Background Therapy) for >=3 Months;
Description: Participants from study MHE100185 who completed the 9 months treatment period and achieved a level of <=10 mg of prednisone at study end and participants who withdrew from the study early who were at a prednisone dose level <=10 mg were analyzed. Duration of doses <= 10 mg were determined by examining changes in the prednisone dosing or allowable alternative corticosteroid medication (prednisone equivalents). Start and stop dates of other HES medications were checked to ensure that they did not overlap with the steroid dosing dates. If overlap occurred, then the number of days <=10 mg during this overlap was considered as zero and the cumulative days reset to zero, as the endpoint was assessing prednisone dose as sole background therapy. The dosing criteria for this endpoint was considered as achieved if the duration of dosing was minimum of 84 days (3months).
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants who entered Stage 2 from study MHE100185 with a prednisone level of <=10 mg prednisone were analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 48
Participants | 43

8. Secondary Outcome: For Those Participants Who Entered Stage 1 From Study MHE100185 With >10 mg Prednisone: Number of Participants Achieving a Prednisone Dose <=10 mg (as Sole Background Therapy) for>=3 Months
Description: Participants from study MHE100185 who completed the 9 months treatment period and achieved a level of >10 mg prednisone at the end of the study and participants who withdrew from the study early who were at a prednisone dose level >10 mg were analyzed. Duration of doses <= 10 mg was determined by examining changes in the prednisone dosing or allowable alternative corticosteroid medication (prednisone equivalents). Start and stop dates of other HES medications were checked to ensure that they do not overlap with the steroid dosing dates. If it did, then the number of days <=10 mg during this overlap was considered as zero and the cumulative days reset to zero, as the endpoint was assessing prednisone dose as sole background therapy. The dosing criteria for this endpoint was considered as achieved if the duration of dosing was minimum of 84 days (3months)
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants who entered Stage 1 from study MHE100185 with >10 mg prednisone were analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 30
Participants | 22

9. Secondary Outcome: Blood Eosinophil Count (With Consideration of the HES Background Therapy) During Stages 1-3
Description: Mean blood eosinophil counts were summarized over time taking into account the effect of HES background therapy. Eosinophil count observations for only those participants taking mepolizumab in conjunction with prednisone or as monotherapy were included.
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Cell/uL
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Cell/uL
  MHE100185 Baseline; n=78 | 456.2 (713.81)
  MHE100901 Baseline, n=65 | 467.2 (719.66)
  Week 12; n= 69 | 176.4 (228.41)
  Week 24; n= 68 | 272.6 (499.78)
  Week 48; n= 59 | 163.1 (146.64)
  Week 72; n=49 | 237.3 (358.36)
  Week 96; n=43 | 272.8 (485.06)
  Week 120; n=40 | 174.3 (172.58)
  Week 144; n=36 | 291.4 (546.03)
  Week 168; n=33 | 210.6 (283.35)
  Week 192; n=27 | 208.5 (249.01)
  Week 216; n=23 | 274.8 (337.50)
  Week 240; n=21 | 138.1 (138.08)
  Week 264; n=9 | 466.7 (533.99)
  Week 288; n=2 | 350.0 (212.13)

10. Secondary Outcome: Number of Participants by Dosing Frequency Groups (Defined as Two Week Dosing Ranges Greater Than a 4 Week Interval) at the End of Stage 2
Description: The number of participants at the end of Stage 2 with study medication dosing frequencies of 4 weeks, 5-6 weeks, 7-8 weeks, 9-10 weeks, 11-12 weeks, 13-16 weeks, 17-20 weeks, 21-24 weeks and >24 weeks were summarized. The first infusion date in Stage 3 and the last infusion date in Stage 2 were used to calculate the dosing frequency.
Time Frame: up to approximately 6 years
Population: ITT Population. Only those participants available at end of Stage 2 were included.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 59
Participants
  <4 Weeks | 1
  4 Weeks | 5
  5 to 6 Weeks | 6
  7 to 8 Weeks | 4
  9 to 10 Weeks | 5
  11 to 12 Weeks | 8
  13 to 16 Weeks | 12
  17 to 20 Weeks | 8
  21 to 24 Weeks | 4
  >24 Weeks | 6

11. Secondary Outcome: Change From Baseline in the Pruritus Visual Analogue Scale (pVAS) 3 Months After the Start of Study MHE100901 and Every 6 Months Thereafter
Description: The pruritus visual analogue scale asks participants to rate the status of their Pruritus based on the severity of their itch. Scores range from 0-100 with 0 = No itch and 100 = Worst imaginable itch. Change from Baseline in pVAS score is the difference between the pVAS score at the time point being considered to the MHE100901 Baseline score.
Time Frame: Baseline and up to approximately 6 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 73
Scores on the scale
  Week 12; n= 58 | -6.8 (20.01)
  Week 24; n= 51 | -4.5 (17.49)
  Week 48; n= 46 | -5.1 (26.19)
  Week 72; n=39 | -0.1 (20.77)
  Week 96; n=41 | 1.0 (27.63)
  Week 120; n=38 | -0.3 (17.84)
  Week 144; n=32 | -2.8 (18.68)
  Week 168; n=33 | -4.9 (26.55)
  Week 192; n=30 | -1.2 (21.54)
  Week 216; n=21 | -0.8 (13.99)
  Week 240; n=17 | 4.4 (12.33)
  Week 264; n=7 | 2.7 (13.14)
  Week 288; n=2 | 39.5 (54.45)

12. Secondary Outcome: Change From Baseline in Erythema/Edema Score 3 Months After the Start of Study MHE100901 and Every 6 Months Thereafter
Description: The erythema subscale score and edema subscale score are each graded on a 0-3 scale, with 0 = absent , 1 = mild, 2 = moderate, 3 = severe. The total score ranged from 0 to 6, with higher scores indicative of more severe Erythema/Edema. The total score was obtained by summing together the responses for each of the two subscale items. Change from Baseline in erythema/edema total score is the difference between erythema/edema total score at the time point being analyzed to the MHE100901 Baseline score..
Time Frame: Baseline and up to approximately 6 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 78
Scores on a scale
  Week 12; n= 59 | 0.0 (1.07)
  Week 24; n= 54 | 0.0 (1.00)
  Week 48; n= 36 | 0.0 (1.13)
  Week 72; n=38 | 0.2 (0.98)
  Week 96; n=21 | -0.1 (1.01)
  Week 120; n=11 | -0.2 (0.60)
  Week 144; n=9 | -0.2 (0.67)
  Week 168; n=6 | 0.5 (1.05)
  Week 192; n=4 | 0.8 (0.96)
  Week 216; n=4 | 0.3 (1.26)
  Week 240; n=11 | 0.3 (0.65)
  Week 264; n=8 | 0.0 (0.00)
  Week 288; n=3 | -1.0 (1.00)

13. Secondary Outcome: Change From Baseline in Quality of Life (QoL) and Current Health Status: Physical Summary Score of the Study Short Form Health Survey (SF-12) 3 Months After the Start of Study MHE100901 and Every 6 Months Thereafter
Description: The SF-12v2 is the 12 item abbreviated form of SF-36v2 survey . It provides information about how participants feel, and how well they have been able to perform their usual activities, over the past 4 weeks. SF-12v2 questions make up 8 scales: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health . Transformed physical component summary score (PCS-12) is derived using all the 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning. Change from Baseline in scale or summary measure score is the difference between the score at the time point being analyzed to Baseline.
Time Frame: Baseline and up to approximately 6 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 75
Scores on the scale
  Week 12; n= 64 | -2.0 (8.25)
  Week 36; n= 50 | -1.4 (8.76)
  Week 60; n=48 | -1.1 (8.91)
  Week 84; n=47 | -0.8 (8.43)
  Week 108; n=39 | -1.0 (8.23)
  Week 132; n=37 | -1.3 (8.33)
  Week 156; n=41 | -1.1 (8.66)
  Week 180; n=45 | -2.1 (8.10)
  Week 204; n=43 | -2.2 (10.02)
  Week 228; n=44 | -0.1 (9.41)
  Week 252; n=24 | -1.3 (9.60)
  Week 276; n=12 | -1.4 (10.76)

14. Secondary Outcome: Change From Baseline in QoL and Current Health Status: Mental Summary Score of the SF12 3 Months After the Start of Study MHE100901 and Every 6 Months Thereafter
Description: The SF-12v2 is the 12 item abbreviated form of SF-36v2 survey developed by the Medical Outcomes Trust and QualityMetric Incorporated. It provides information about how participants feel, and how well they have been able to perform their usual activities, over the past 4 weeks. SF-12v2 scale questions make up 8 scales: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health are for mental component summary. Transformed mental component summary score (MCS-12) is derived using all the 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning. Change from Baseline in scale or summary measure score is the difference between the score at the time point being analyzed to Baseline.
Time Frame: Baseline and up to approximately 6 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 75
Scores on a scale
  Week 12; n= 64 | 2.8 (8.46)
  Week 36; n= 50 | 1.6 (10.75)
  Week 60; n=48 | 2.8 (10.34)
  Week 84; n=47 | 1.5 (8.46)
  Week 108; n=39 | 2.9 (11.02)
  Week 132; n=37 | 5.3 (10.20)
  Week 156; n=41 | 2.1 (10.82)
  Week 180; n=45 | 2.7 (11.95)
  Week 204; n=43 | 1.9 (11.54)
  Week 228; n=44 | 1.8 (11.43)
  Week 252; n=24 | 0.6 (12.13)
  Week 276; n=12 | 3.3 (12.44)

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from from the first dose of study medication up to 7 days after the last dose (up to approximately 6 years).
Description: SAEs and non-serious AEs were collected in members of the Intent to treat (ITT)population, comprised of all enrolled participants who received at least one dose of mepolizumab in this study
Arm/Group | Mepolizumab 750 mg
Serious Adverse Events (participants affected / at risk) | 40/78
Other Adverse Events (participants affected / at risk) | 72/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 750 mg (N=78)
Pneumonia (Infections and infestations) | 4
Acquired immunodeficiency syndrome (Infections and infestations) | 1
Bronchiectasis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis clostridial (Infections and infestations) | 1
HIV infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Pyrexia (General disorders) | 3
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Multi-organ failure (General disorders) | 1
Sudden death (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Motor neurone disease (Nervous system disorders) | 1
Myelitis transverse (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Radiculitis brachial (Nervous system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arterial occlusive disease (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Temporal arteritis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Infections and infestations) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Eosinophilic cellulitis (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Swelling face (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholangitis sclerosing (Hepatobiliary disorders) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hepatic enzyme increased (Investigations) | 1
T-lymphocyte count increased (Investigations) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Self-injurious ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 750 mg (N=78)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 22
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 22
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 21
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 18
Rhinitis (Infections and infestations) | 9
Ear infection (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 6
Cystitis (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 5
Localised infection (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 5
Fungal infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Fatigue (General disorders) | 23
Pyrexia (General disorders) | 14
Influenza like illness (General disorders) | 10
Pain (General disorders) | 10
Oedema peripheral (General disorders) | 9
Chest pain (General disorders) | 8
Oedema (General disorders) | 7
Asthenia (General disorders) | 5
Local swelling (General disorders) | 4
Nausea (Gastrointestinal disorders) | 18
Abdominal pain (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 10
Abdominal pain upper (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Abdominal discomfort (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 4
Oesophagitis (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Asthma (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 15
Urticaria (Skin and subcutaneous tissue disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 5
Headache (Nervous system disorders) | 23
Hypoaesthesia (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 6
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 5
Weight decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 7
Contusion (Injury, poisoning and procedural complications) | 6
Palpitations (Cardiac disorders) | 5
Vision blurred (Eye disorders) | 4
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.